



Medical Unit: Subdirección de Enseñanza e Investigación C.M.N. "November 20"

# IDENTIFICATION OF BIOMARKERS DERIVED FROM ADIPOSE TISSUE WITH POTENTIAL UTILITY IN THE DIAGNOSIS AND PROGNOSIS OF CARDIOVASCULAR RISK OF OBESE PATIENT

DR. JUAN ANTONIO SUAREZ CUENCA, DR. MOISES ORTIZ FERNANDEZ, DRA. JULITA OROZCO VÁZQUEZ, DR. MARIO OSORIO VALERO and DR. ALBERTO MELCHOR LOPEZ.

#### Background

Obesity is a nutritional disorder that is considered a risk factor for several metabolic abnormalities, such as insulin resistance, Diabetes Mellitus type 2 (DM2), NAFLD, endothelial dysfunction, cardiovascular risk and is associated with high morbidity and mortality.

According to the panel of experts from the National Heart and Lung Institute of the United States, "obesity is a chronic disease that results from the interaction of the genotype and the environment." In 1997, the World Health Organization defined obesity as "an excess of fat that accumulates in such an amount that health can be adversely affected." In Mexico, obesity represents a priority problem for public health, since its high frequency places the country in second place of prevalence worldwide.

A scale to classify obesity is the body mass index (BMI), in which the obese subject is one with a BMI  $\geq$  30kg / m2 and subdivided into 3 classes (Table 1).

| Table 1. Body Weight Classification According to the BMI in Adults | |
|---|---|
| | BMI |
| Normal | 18.5-24.9 kg / m2 |
| Obese Grade 1 | 30-34.9 kg / m2 |
| Obese Grade 2 | 35.0 -39.9 kg / m2 |
| Obese Grade 3 | ≥40 kg / m2 |

### **Morbid Obesity**

Morbid obesity refers to an extreme degree of obesity, which affects basic physiological functions and is related to specific risks (Table 2). It has been estimated that a morbid obese man reduces his life expectancy by up to 22% compared to an individual of normal weight.

| Table 2. Impact on the long-term health of morbid obesity |
|----------------------------------------------------------------------|
| Decreased life expectancy |
| Dyslipidemia |
| Decrease in the quality of life of economic and social opportunities |
| Obstructive sleep apnea |
| Cardiovascular diseases |
| Gastroesophageal reflux disease |
| DM2 |
| Cancer |
| Depression |
| Osteoarthritis |
| Hypertension |
| Kidney failure |

#### **Bariatric Surgery**

Bariatric surgery not only induces weight loss, but also significantly improves the covariabilities associated with morbid obesity in those patients accepted. Clinical trials and observational studies have shown that bariatric surgery can prolong survival in patients with extreme obesity. In fact, the National Institutes of Health of the United States recommend bariatric surgery that should be presented with BMI> 40 kg / m2 or> 35 kg / m2 concomitant related to obesity.

Surgeries to reduce food intake reduce the amount of oral intake through a bag that limits the passage of food. It has also been proposed that a) it would induce a sense of emergence or suppression of appetite as a mechanism in weight loss; b) compress the vagus nerve; c) decreased the secretion of gastrointestinal hormones, such as ghrelin or peptide YY. The surgeries that are included in this type are the adjustable gastric band and sleeve gastrectomy.

Hybrid procedures are represented by the gastric Roux-en-Y derivation (DYRG), which involves reducing the size of the stomach by 15 ml by resecting the upper stomach portion and anastomosing it to the small intestine. The stomach remains viable but the

food is derived from the small intestine and the remaining stomach has a lower capacity; the duodenum does not absorb the macronutrients responsible for post-prandial hormonal responses.

Appetite reduction can be partially explained by the YY principle and the glucagon-like principle1-3 The duodenum bypass also contributes to decrease the absorption of iron and calcium, requiring its supplementation4. The biliopancreatic diversion (BPD) involves the resection of the upper 2/3 of the stomach, leaving a stomach capacity of 250 ml, disconnecting half of the jejunum and ileum from the alimentary tract and reconnecting it to the terminal ileum. With the delay in the action of the digestive enzymes within the alimentary tract, most of the fat and a significant fraction of the proteins is excreted as a result of the decrease in its ingestion. There is a dramatic loss in weight, but certain micronutrients are not absorbed, so supplements are required. There is a modification of DBP, called "switch" DBP, which consists of a sleeve gastrectomy with a less dramatic intestinal derivation. The difference lies in the preservation of the pylorus, which leads to fewer complications.

Postoperative mortality at 30 days ranges from 0.1% to 2% 5-7 and depends on the complexity of the operation, the co-morbidities of the patient, the experience of the surgeon and the hospital institution. The patient with morbid obesity can be complicated early by thromboembolism (1%), respiratory failure (<1%) hemorrhage (1%), peritonitis (1%) and / or wound infection (2%). Laparoscopy has been useful in reducing these rates. On the other hand, late complications include obstruction, ulcerations, hypoglycemia, steatorrhea, and bacterial overgrowth. Dietary modification and antibiotics can help control the severity of these side effects.

Bariatric Surgery - Metabolic and Cardiovascular Benefits

Bariatric surgery offers sustained weight loss. On average, time loses 50% of the weight of the 5 years, although this depends on the type, aggressiveness and complexity of the surgery.

Effect on DM2. Up to 50% -60% of patients with DM2 are known as morbidly obese. The most relevant clinical impact of surgically induced weight loss is the ability to completely reverse DM2 in a large percentage of patients. In a long-term study of surgical and conventional therapy, DM2 was reversed in 21% of the control group and in 72% of the study group after 2 years of follow-up.55 At 10 years of follow-up, DM2 it could be reversed in 13% of the control group and in 36% of the group with surgery. The odds ratio on recovery of DM2 with surgery at 2 years was 8.42 (95% confidence interval, 5.68 to 12.5) and at 10 years it was 3.45 (95% interval)

#### JUSTIFICATION

Bariatric surgery induces a significant reduction in the co-morbidities associated with obesity, such as DM2, dyslipidemia, liver disease, arterial hypertension, obstructive sleep apnea and cardiovascular risk. However, this does not happen in all obese patients, even when there is a reduction in weight.

It is known that adipose tissue participates actively in the synthesis of cytokines and its constitutive role in metabolic phenotypes has been suggested. It is possible that the

intrinsic mechanisms of adipose tissue participate in several benefits observed in morbidly obese patients who undergo anti-obesity surgery. Therefore, this study explores the participation of adipose tissue, as an active component, that can define metabolic phenotypes linked to the modification of cardiovascular risk after bariatric surgery.

#### **HYPOTHESIS**

- H1 Metabolic phenotypes based on basic mechanisms of adipose tissue are associated to the cardiovascular risk modification after bariatric surgery.
- H0. Metabolic phenotypes based on basic mechanisms of adipose tissue are NOT associated to the cardiovascular risk modification after bariatric surgery.

#### **GENERAL OBJETIVE**

To evaluate the association of the cardiovascular benefit of the obese patient after bariatric surgery with the basic mechanisms of adipose tissue (metabolic profile)

#### **SPECIFIC OBJECTIVES**

- a) Characterize the basal (pre-surgical) metabolic profile of adipose tissue.
- b) Evaluate post-surgical modification of cardiovascular prognosis
- c) Determine the association of the cardiovascular prognosis modification (risk subgroups) with the basal metabolic profile.

#### **DESIGN**

This is an OBSERVATIONAL study, of a prospective cohort follow-up. We will study morbidly obese patients who undergo bariatric surgery (this is not a proposal of the present protocol, it is routinely done as a treatment for morbid obesity in the CMN "20 de Noviembre", ISSSTE, and it would also be carried out although the patient does not participate in this study). It was considered that the independent variable is the change in cardiovascular risk after bariatric surgery and the dependent variable is the basal metabolic profile of adipose tissue. This order of variables was decided by methodological strategy, since it will be more convenient to determine and stratify based on the change in cardiovascular risk, than based on the basal metabolic profile of adipose tissue.

$$n = \frac{(Z^{\alpha/2})^2 (p(1-p))}{d^2}$$

where:

n = sample size.  $Z^{a/2} = Z^{-1}$  value of the alpha error with a confidence of 95%, assigning alpha = 0.05  $p = Z^{a/2}$  Expected population prevalence for the event under study (according to previous reports).  $z = Z^{a/2} = Z^{-1}$ 

=difference between the expected population prevalence value and the acceptable error. Considering the average difference in the modification of the basic mechanisms in adipose tissue associated with metabolic risk in similar studies

$$(1.96)^2 (0.20 (1-0.20))$$
 0.614  
 $n =$   $n =$   $= 36.3$   
 $(0.13)^2$  0.0169

Additionally, for reasons of comparison and standardization of results, a C group would be considered: 10 non-obese patients undergoing non-bariatric surgery.

#### Definition of the observation units.

Patients with morbid obesity subjected to bariatric surgery, with significant modification of cardiovascular risk in the postoperative period.

#### **Definition of the control group**

Due to the observational design of the before-after evaluation (of bariatric surgery), the morbidly obese patient in the pre-surgical baseline is his own reference ("control") for the postoperative period. It is also considered non-obese subjects subjected to abdominal surgery eg. Hernioplasty, fundoplication etc. to know the "nomal" metabolic profile of adipose tissue.

#### Inclusion criteria

- · Men and women.
- Over 18 years.
- With morbid obesity and candidates for bariatric surgery, under the routine of the treating service.
- Signature of acceptance of your participation, through informed consent.

#### **Exclusion criteria.**

- Medication with potential effect on fatty tissue or cardiovascular risk in the last month.
- Serious infections in the last month.
- Clinically unstable conditions.

#### Elimination criteria.

- Desire not to continue in the study
- Samples or insufficient information for an adequate analysis.

## Definition of variables and units of measurement.

| Definition of variables and units of measurement. | | | |
|---|---|---|---|
| Variable | Dependent /<br>Independent | Туре | Units of measurement |
| Total body fat, visceral and subcutaneous | Dependent | Discontinuous<br>Quantitative | Percentage |
| Serum markers of inflammation PCR and IL- | Dependent | Quantitative continuous | μUI / dL |
| Serum adipokines: leptin and adiponectin | Dependent | Quantitative continuous | μUI / dL |
| Differentiation and hypertrophy of adipocytes and angiogenesis | Dependent | Qualitative dichotomous | Present or absent |
| Pro-inflammatory markers at tissue level | Dependent | Qualitative dichotomous | Present or absent |
| Oxidative stress and tissue endoplasmic reticulum | Dependent | Qualitative dichotomous | Present or absent |
| Insulin sensitivity | Dependent | Qualitative dichotomous | Sensitive or not sensitive |
| НОМА | Dependent | Qualitative dichotomous | Higher or lower than 15 |
| Prognostic scales<br>mortality due to<br>independent<br>cardiovascular cause | Independent | Quantitative<br>discontinuous | Own rating |
| Flow mediaded dilatation | Independent | Quantitative discontinuous | Percentage |
| Carotid intima media thickness | Independent | Quantitative discontinuous | Millimeters |

# Selection of sources, methods, techniques and procedures for collecting information

With the acceptance of the Institutional Ethics, Research and Biosafety Committees, patients will be invited and included according to the selection criteria.

Prior signature of informed consent, will include patients with morbid obesity, candidates for bariatric surgery and without additional modifiers of adipose tissue metabolism. Patients will be chosen in accordance with the criteria of the Bariatric Surgery Service, without modifying the routine procedures performed in this service.

At the same time, a group of non-obese patients (obesity comparison group) scheduled and undergoing non-bariatric abdominal surgery (hernioplasty, cholecystectomy, appendectomy, etc.) will be included. In all groups, total body fat, subcutaneous and visceral fat will be determined non-invasively by computed tomography, with the support of the Department of Imaging (Dr. Julita Orozco and Dr. Mario Osorio) as described below:

#### TOMOGRAPHIC MEASUREMENT OF SUBCUTANEOUS AND VISCERAL GREASE

#### Subcutaneous fat:

The thickness of adipose tissue will be measured, in the abdominal thickest site, at the level of the umbilical scar, with references from the skin to the muscular layer, either in vertical measurement (antero-posterior) or in lateral measurement.

#### Visceral fat:

Epicardial fat: The thickness of the adipose tissue will be measured epicardial level, in the thickest site.

#### Preperitoneal fat:

The thickness of adipose tissue will be measured,

level of the umbilical scar; from the muscular layer (vertical measurement or ant-post) to the first visceral structure.

#### Perirenal fat:

The thickness of adipose tissue will be measured perirenal, in the thickest site.

During the surgical act, a sample of 1-2 cubic cm of visceral and subcutaneous adipose tissue will be taken, in all groups, considering all aspects of patient Ethics and Biosafety described in the respective sections of this project. In patients with laboratorial evidence and image of progression to NAFLD, a sample of 1-2 cubic cm of liver tissue will be taken, in accordance with international guidelines for diagnosis and treatment, and with the study protocol established by the service. It will be guaranteed that the taking of biopsies will not affect the course of the surgery. The biological samples acquired will be properly identified, contained and stored for a maximum period of 1 year. Analysis and determinations will be made according to good laboratory practices. Subsequently, they will be treated and disposed of in appropriate bags for disposal. To comply with the provisions of section 6 of NOM-087-ECOL-SSA1-2002 Biological-Infectious Waste.

To study the characteristics of each metabolic profile, the following variables will be analyzed:

- a) Adipose tissue (visceral and subcutaneous) where the degree of differentiation and hypertrophy of adipocytes and angiogenesis will be determined by morphometric methods of histopathology; as well as markers of inflammation, oxidative stress, endoplasmic reticulum stress and adipose tissue dysfunction through immunohistochemistry and in vitro tests on isolated adipocytes.
- b) Liver tissue the degree of steatosis, steatohepatitis and fibrogenesis, considered as clinical progression of metabolic damage, will be determined.
- c) Serum level, inflammation markers (TNFa, CRP and IL-6) and adipokines (leptin, adiponectin, resistin) will be determined by ELISA.

Finally, in all groups, follow-up variables related to post-surgical modification of cardiovascular risk will be determined; through:

Prognostic scales of cardiovascular mortality: They will be determined by Drs. Moises Ortíz and Juan Suárez Cuenca, based on probability calculation with variables such as age, gender, co-morbidities, etc. using Framingham or SCORE scales. Place: Clinical Research Division, CMN "November 20", ISSSTE.

Determination of serum markers of endothelial dysfunction and ankle / arm index. They will be determined by Dr. Juan Suárez Cuenca and associated researchers, using commercially available ELISA kits and direct determination of systolic pressure in the ankle and arm, with the help of Doppler scan type Doptone, respectively. Place: Biomedical Research Laboratory and Clinical Research Division, CMN "November 20", ISSSTE.

Determination of subclinical atherogenesis (thickness of the carotid intima media). It will be determined by the Department of Imaging, with the support of Dr. Toriz. The Doppler transducer will be placed in the neck and the common carotid artery will be located, then the thickness of the intimal vascular mean will be determined 1 cm from the carotid bifurcation. The determination will be made by two observers to estimate the inter-observer correlation. Place: Department of Imaging, CMN "November 20", ISSSTE.

The determination of these variables of cardiovascular risk modification will be determined basally and periodically at 3, 6 and 9 months after bariatric surgery, in all groups.

Definition of the processing plan and presentation of the information

Data analysis will be done through descriptive statistics applied to demographic variables, and inferential statistics, which will include difference of averages, correlation, strength of association and relative risk, as well as multivariate logistic regression analysis to evaluate independent associations. With the variables most associated with the modification of cardiovascular risk, a metabolic profile will be established as a predictive model of the greatest cardiovascular benefit after bariatric surgery. Statistical significance will be considered with p <0.05

#### **ETHICAL CONSIDERATIONS**

This study is considered as minimal risk. Bariatric surgery (this procedure is not a proposal of the present protocol, it is routinely done as a treatment for morbid obesity in the CMN "20 de Noviembre", ISSSTE and would also be done if the patient does not participate in the study) will be performed according to the routine procedures of the Department of Bariatric Surgery. The project complies with the guidelines and recommendation of the Declaration of Helsinki. The protocol will be submitted to the Ethics and Institutional Research Committee. All patients will be asked to read and sign informed consent.

#### **BIOSECURITY CONSIDERATIONS.**

Bariatric surgery procedures are not part of this investigation. In any case, it is emphasized that this project does not alter the surgical procedure and routine biosecurity measures, which are based on the best clinical practice and international recommendations (Neff KJ, le Roux CW, Bariatric surgery: a best practice article. Pathol 2013; 66: 90-8). Sampling during surgery will be done in accordance with the Regulation of the General Health Law on Health Research, respecting aspects of taking the appropriate measures to avoid any risk or damage to research subjects (includes adequate preoperative assessment). , biosecurity measures typical of an operating room and sampling by an experienced surgeon). In any case, the privacy of the individual subject of the investigation will be protected, and it will be sought to limit the likelihood that the subject will suffer any harm as a result of the study.

The biological samples acquired will be properly identified, contained and stored for a maximum period of 1 year. Your analysis and determinations will be made according to good laboratory practices. Subsequently, they will be treated and disposed of in appropriate bags for disposal. To comply with the provisions of section 6 of NOM-087-ECOL-SSA1-2002 Biological-Infectious Waste.

The research is considered to be of minimal risk, since it is a common procedure with obtaining a minimum sample of visceral and subcutaneous adipose tissue. Likewise, the principal investigator will suspend the investigation upon noticing any risk or damage to the health of the subject in whom the investigation is carried out. All participants will read, understand and sign an informed consent.

#### **BIBLIOGRAPHY**

- 1. TROY S, SOTY M, RIBEIRO L, MIGRENNE S, FIORAMONTI X, PILLOT B, FAUVEAU V, AUBERT R, VIOLLET B, FORETZ M, LECLERC J, DUCHAMPT A, ZITOUN C, THORENS B, MAGNAN C, MITHIEUX G, ANDREELLI F. INTESTINAL GLUCONEOGENESIS IS A KEY FACTOR FOR EARLY METABOLIC CHANGES AFTER GASTRIC BYPASS BUT NOT AFTER GASTRIC LAP-BAND IN MICE. CELL METAB. 2008;8:201–211.
- LAFERRERE B, HESHKA S, WANG K, KHAN Y, MCGINTY J, TEIXEIRA J, HART AB, OLIVAN B. INCRETIN LEVELS AND EFFECT ARE MARKEDLY ENHANCED 1 MONTH AFTER ROUX-EN-Y GASTRIC BYPASS SURGERY IN OBESE PATIENTS WITH TYPE 2 DIABETES. DIABETES CARE. 2007;30:1709 –1716.
- 3. YE ROUX CW, WELBOURN R, WERLING M, OSBORNE A, KOKKINOS A, LAURENIUS A, LONROTH H, FANDRIKS L, GHATEI MA, BLOOM SR, OLBERS T. GUT HORMONES AS MEDIATORS OF APPETITE AND WEIGHT LOSS AFTER ROUX-EN-Y GASTRIC BYPASS. ANN SURG. 2007;246:780 –785.
- 4. GUIDELINES FOR REPORTING RESULTS IN BARIATRIC SURGERY: STANDARDS COMMITTEE, AMERICAN SOCIETY FOR BARIATRIC SURGERY. OBES SURG. 1997;7:521–522.
- 5. BUCHWALD H, ESTOK R, FAHRBACH K, BANEL D, SLEDGE I. TRENDS IN MORTALITY IN BARIATRIC SURGERY: A SYSTEMATIC REVIEW AND META-ANALYSIS. SURGERY. 2007; 142:621–32.
- 6. BUCHWALD H, AVIDOR Y, BRAUNWALD E, JENSEN MD, PORIES W, FAHRBACH K, SCHOELLES K. BARIATRIC SURGERY: A SYSTEMATIC REVIEW AND META-ANALYSIS. JAMA. 2004;292:1724 –1737.
- 7. BUCHWALD H. BARIATRIC SURGERY FOR MORBID OBESITY: HEALTH IMPLICATIONS FOR PATIENTS, HEALTH PROFESSIONALS, AND THIRD-PARTY PAYERS. J AM COLL SURG. 2005;200:593–604.
- 8. HESS DS; 2004 ABS CONSENSUS CONFERENCE. BILIOPANCREATIC DIVERSION WITH DUODENAL SWITCH. SURG OBES RELAT DIS. 2005;1:329 333.
- 9. LEIBSON CL, WILLIAMSON DF, MELTON LJ 3RD, PALUMBO PJ, SMITH SA, RANSOM JE, SCHILLING PL, NARAYAN KM. TEMPORAL TRENDS IN BMI AMONG ADULTS WITH DIABETES. DIABETES CARE. 2001;24:1584.
- 10. SJOSTROM L, LINDROOS AK, PELTONEN M, TORGERSON J, BOUCHARD C, CARLSSON B, DAHLGREN S, LARSSON B, NARBRO K, SJOSTROM CD, SULLIVAN M, WEDEL H; SWEDISH OBESE SUBJECTS STUDY SCIENTIFIC GROUP. LIFESTYLE, DIABETES, AND CARDIOVASCULAR RISK FACTORS 10 YEARS AFTER BARIATRIC SURGERY.N ENGL J MED. 2004: 351:2683–2693.

- 11. SCHERNTHANER G, MORTON JM. BARIATRIC SURGERY IN PATIENTS WITH MORBIDOBESITY AND TYPE 2 DIABETES. DIABETES CARE. 2008;31(SUPPL 2):S297–S302.
- 12. ISBELL JM, TAMBOLI RA, HANSEN EN, SALIBA J, DUNN JP, PHILLIPS SE, MARKS-SHULMAN PA, ABUMRAD NN. THE IMPORTANCE OF CALORIC RESTRICTION IN THE EARLY IMPROVEMENTS IN INSULIN SENSITIVITY AFTER ROUX-EN-Y GASTRIC BYPASS SURGERY. DIABETES CARE. 2010;33:1438 1442.
- 13. LAFERRERE B, TEIXEIRA J, MCGINTY J, TRAN H, EGGER JR, COLARUSSO A, KOVACK B, BAWA B, KOSHY N, LEE H, YAPP K, OLIVAN B. EFFECT OF WEIGHT LOSS BY GASTRIC BYPASS SURGERY VERSUS HYPOCALORIC DIET ON GLUCOSE AND INCRETIN LEVELS IN PATIENTS WITH TYPE 2 DIABETES. J CLIN ENDOCRINOL METAB. 2008;93:2479 –2485.
- 14. BOSE M, OLIVAN B, TEIXEIRA J, PI-SUNYER FX, LAFERRERE B. DO INCRETINS PLAY A ROLE IN THE REMISSION OF TYPE 2 DIABETES AFTER GASTRIC BYPASS SURGERY: WHAT ARE THE EVIDENCE? OBES SURG. 2009;19:217–229.
- 15. BROLIN RE, KENLER HA, WILSON AC, KUO PT, CODY RP. SERUM LIPIDS AFTER GASTRIC BYPASS SURGERY FOR MORBID OBESITY. INT J OBES. 1990;14: 939–950.
- 16. BROLIN RE, BRADLEY LJ, WILSON AC, CODY RP. LIPID RISK PROFILE ANDVWEIGHT STABILITY AFTER GASTRIC RESTRICTIVE OPERATIONS FOR MORBID OBESITY. J GASTROINTEST SURG. 2000;4:464–469.
- 17. NGUYEN NT, VARELA E, SABIO A, TRAN CL, STAMOS M, WILSON SE. RESOLUTION OF HYPERLIPIDEMIA AFTER LAPAROSCOPIC ROUX-EN-Y GASTRIC BYPASS. J AM COLL SURG. 2006;203:24 –29.
- 18. DHABUWALA A, CANNAN RJ, STUBBS RS. IMPROVEMENT IN CO-MORBIDITIES FOLLOWING WEIGHT LOSS FROM GASTRIC BYPASS SURGERY. OBES SURG. 2000;10: 428–435.
- 19. GLEYSTEEN JJ, BARBORIAK JJ, SASSE EA. SUSTAINED CORONARY-RISK-FACTOR REDUCTION AFTER GASTRIC BYPASS FOR MORBID OBESITY. AM J CLIN NUTR. 1990;51:774 –778.
- 20. GLEYSTEEN JJ. RESULTS OF SURGERY: LONG-TERM EFFECTS ON HYPERLIPIDEMIA. AM J CLIN NUTR. 1992;55(SUPPL):591S-593S.

- 21. COWAN GS JR, BUFFINGTON CK. SIGNIFICANT CHANGES IN BLOOD PRESSURE, GLUCOSE, AND LIPIDS WITH GASTRIC BYPASS SURGERY. WORLD J SURG. 1998; 22: 987–992.
- 22. DIXON JB, O'BRIEN PE. LIPID PROFILE IN THE SEVERELY OBESE: CHANGES WITH WEIGHT LOSS AFTER LAP-BAND SURGERY. OBES RES. 2002;10:903–910.
- 23. HANUSCH-ENSERER U, CAUZA E, SPAK M, ENDLER G, DUNKY A, TURA A, WAGNER O, ROSEN HR, PACINI G, PRAGER R. IMPROVEMENT OF INSULIN RESISTANCE AND EARLY ATHEROSCLEROSIS IN PATIENTS AFTER GASTRIC BANDING. OBES RES. 2004;12:284 –291.
- 24. DESPRES JP, POIRIER P, BERGERON J, TREMBLAY A, LEMIEUX I, ALMÉRAS N. FROM INDIVIDUAL RISK FACTORS AND THE METABOLIC SYNDROME TO GLOBAL CARDIOMETABOLIC RISK. EUR HEART J. 2008;10(SUPPL B):B24–B33.
- 25. MATHIEU P, POIRIER P, PIBAROT P, LEMIEUX I, DESPRES JP. VISCERAL OBESITY: THE LINK AMONG INFLAMMATION, HYPERTENSION, AND CARDIOVASCULAR DISEASE. HYPERTENSION. 2009;53:577–584.
- 26. AIGNER F, PATSCH JR. MARKERS OF CHRONIC INFLAMMATION AND OBESITY: A PROSPECTIVE STUDY ON THE REVERSIBILITY OF THIS ASSOCIATION IN MIDDLE-AGED WOMEN UNDERGOING WEIGHT LOSS BY SURGICAL INTERVENTION. INT J OBES RELAT METAB DISORD. 2002;26:659– 662.
- 27. KOPP HP, KOPP CW, FESTA A, KRZYZANOWSKA K, KRIWANEK S, MINAR E, ROKA R, SCHERNTHANER G. IMPACT OF WEIGHT LOSS ON INFLAMMATORY PROTEINS AND THEIR ASSOCIATION WITH THE INSULIN RESISTANCE SYNDROME IN MORBIDLY OBESE PATIENTS. ARTERIOSCLER THROMB VASC BIOL. 2003;23: 1042–1047.
- 28. HANUSCH-ENSERER U, CAUZA E, SPAK M, DUNKY A, ROSEN HR, WOLF H, PRAGER R, EIBL MM. ACUTE-PHASE RESPONSE AND IMMUNOLOGICAL MARKERS IN MORBID OBESE PATIENTS AND PATIENTS FOLLOWING ADJUSTABLE GASTRIC BANDING. INT J OBES RELAT METAB DISORD. 2003;27:355–361.
- 29. VAZQUEZ LA, PAZOS F, BERRAZUETA JR, FERNANDEZ-ESCALANTE C, GARCIA-UNZUETA MT, FREIJANES J, AMADO JA. EFFECTS OF CHANGES IN BODY WEIGHT AND INSULIN RESISTANCE ON INFLAMMATION AND ENDOTHELIAL FUNCTION IN MORBID OBESITY AFTER BARIATRIC SURGERY. J CLIN ENDOCRINOL METAB. 2005; 90:316 –322.

- 30. ZAGORSKI SM, PAPA NN, CHUNG MH. THE EFFECT OF WEIGHT LOSS AFTER GASTRIC BYPASS ON C-REACTIVE PROTEIN LEVELS. SURG OBES RELAT DIS. 2005; 1:81–85.
- 31. KOPP HP, KRZYZANOWSKA K, MOHLIG M, SPRANGER J, PFEIFFER AF, SCHERNTHANER G. EFFECTS OF MARKED WEIGHT LOSS ON PLASMA LEVELS OF ADIPONECTIN, MARKERS OF CHRONIC SUBCLINICAL INFLAMMATION AND INSULIN RESISTANCE IN MORBIDLY OBESE WOMEN. INT J OBES (LOND). 2005;29:766 –771.
- 32. HOLDSTOCK C, LIND L, ENGSTROM BE, SUNDBOM M, LARSSON A, KARLSSON FA. CRP REDUCTION FOLLOWING GASTRIC BYPASS SURGERY IS MOST PRONOUNCED IN INSULIN-SENSITIVE SUBJECTS. INT J OBES (LOND). 2005;29:1275–1280.
- 33. SERRA A, GRANADA ML, ROMERO R, BAYES B, CANTON A, BONET J, RULL M, ALASTRUE A, FORMIGUERA X. THE EFFECT OF BARIATRIC SURGERY ON ADIPOCYTOKINES, RENAL PARAMETERS AND OTHER CARDIOVASCULAR RISK FACTORS IN SEVERE AND VERY SEVERE OBESITY: 1-YEAR FOLLOW-UP. CLIN NUTR. 2006;25:400–408.
- 34. SCHERNTHANER GH, KOPP HP, KRIWANEK S, KRZYZANOWSKA K, SATLER M, KOPPENSTEINER R, SCHERNTHANER G. EFFECT OF MASSIVE WEIGHT LOSS INDUCED BY BARIATRIC SURGERY ON SERUM LEVELS OF INTERLEUKIN-18 AND MONOCYTECHEMOATTRACTANT- PROTEIN-1 IN MORBID OBESITY. OBES SURG. 2006;16:709–715.
- VILARRASA N, VENDRELL J, SANCHEZ-SANTOS R, BROCH M, MEGIA A, MASDEVALL C, GOMEZ N, SOLER J, PUJOL J, BETTONICA C, ARANDA H, GOMEZ JM.EFFECT OF WEIGHT LOSS INDUCED BY GASTRIC BYPASS ON PROINFLAMMATORY INTERLEUKIN-18, SOLUBLE TUMOUR NECROSIS FACTOR-ALPHA RECEPTORS, C-REACTIVE PROTEIN AND ADIPONECTIN IN MORBIDLY OBESE PATIENTS. CLIN ENDOCRINOL (OXF). 2007;67:679–686.
- 36. MANCO M, FERNANDEZ-REAL JM, EQUITANI F, VENDRELL J, VALERA MORA ME, NANNI G, TONDOLO V, CALVANI M, RICART W, CASTAGNETO M, MINGRONE G. EFFECT OF MASSIVE WEIGHT LOSS ON INFLAMMATORY ADIPOCYTOKINES AND THE INNATE IMMUNE SYSTEM IN MORBIDLY OBESE WOMEN. J CLIN ENDOCRINOL METAB. 2007;92:483–490.
- 37. IANNELLI A, ANTY R, PICHE T, DAHMAN M, GUAL P, TRAN A, GUGENHEIM J. IMPACT OF LAPAROSCOPIC ROUX-EN-Y GASTRIC BYPASS ON METABOLIC SYNDROME, INFLAMMATION, AND INSULIN RESISTANCE IN SUPER VERSUS MORBIDLY OBESE WOMEN. OBES SURG. 2009;19:577–582.

- 38. AGRAWAL V, KRAUSE KR, CHENGELIS DL, ZALESIN KC, ROCHER LL, MCCULLOUGH PA. RELATION BETWEEN DEGREE OF WEIGHT LOSS AFTER BARIATRIC SURGERY AND REDUCTION IN ALBUMINURIA AND C-REACTIVE PROTEIN. SURG OBES RELAT DIS. 2009;5:20 –26.
- 39. KLEIN S, WADDEN T, SUGERMAN HJ. AGA TECHNICAL REVIEW ON OBESITY. GASTROENTEROLOGY. 2002;123:882–932.
- 40. KLEINER DE, BRUNT EM, VAN NATTA M, BEHLING C, CONTOS MJ, CUMMINGS OW, FERRELL LD, LIU YC, TORBENSON MS, UNALP-ARIDA A, YEH M, MCCULLOUGH AJ, SANYAL AJ; NONALCOHOLIC STEATOHEPATITIS CLINICAL RESEARCH NETWORK. DESIGN AND VALIDATION OF A HISTOLOGICAL SCORING SYSTEM FOR NONALCOHOLIC FATTY LIVER DISEASE. HEPATOLOGY. 2005;41: 1313–1321
- 41. KELLEY DE, MOKAN M, SIMONEAU JA, MANDARINO LJ. INTERACTION BETWEEN GLUCOSE AND FREE FATTY ACID METABOLISM IN HUMAN SKELETAL MUSCLE. J CLIN INVEST. 1993;92:91–98.
- 42. FERRANNINI E, BARRETT EJ, BEVILACQUA S, DEFRONZO RA. EFFECT OF FATTY ACIDS ON GLUCOSE PRODUCTION AND UTILIZATION IN MAN. J CLIN INVEST. 1983;72:1737–1747.
- 43. LEWIS GF, UFFELMAN KD, SZETO LW, WELLER B, STEINER G. INTERACTION BETWEEN FREE FATTY ACIDS AND INSULIN IN THE ACUTE CONTROL OF VERY LOW DENSITY LIPOPROTEIN PRODUCTION IN HUMANS. J CLIN INVEST. 1995;95: 158–166.
- 44. SHOELSON SE, GOLDFINE AB. GETTING AWAY FROM GLUCOSE: FANNING THE FLAMES OF OBESITY-INDUCED INFLAMMATION. NAT MED. 2009;15:373–374.
- 45. KRAL JG, THUNG SN, BIRON S, HOULD FS, LEBEL S, MARCEAU S, SIMARD S, MARCEAU P. EFFECTS OF SURGICAL TREATMENT OF THE METABOLIC SYNDROME ON LIVER FIBROSIS AND CIRRHOSIS. SURGERY. 2004;135:48 –58.
- 46. KLEIN S, MITTENDORFER B, EAGON JC, PATTERSON B, GRANT L, FEIRT N, SEKI E, BRENNER D, KORENBLAT K, MCCREA J. GASTRIC BYPASS SURGERY IMPROVES METABOLIC AND HEPATIC ABNORMALITIES ASSOCIATED WITH NONALCOHOLIC FATTY LIVER DISEASE. GASTROENTEROLOGY. 2006; 130:1564 –1572.
- 47. STAMLER R, STAMLER J, RIEDLINGER WF, ALGERA G, ROBERTS RH. WEIGHT AND BLOOD PRESSURE: FINDINGS IN HYPERTENSION SCREENING OF 1 MILLION AMERICANS. JAMA. 1978;240:1607–1610.

- 48. WEYER C, PRATLEY RE, SNITKER S, SPRAUL M, RAVUSSIN E, TATARANNI PA. ETHNIC DIFFERENCES IN INSULINEMIA AND SYMPATHETIC TONE AS LINKS BETWEEN OBESITY AND BLOOD PRESSURE. HYPERTENSION. 2000;36:531–537.
- 49. MASUO K, MIKAMI H, OGIHARA T, TUCK ML. DIFFERENCES IN MECHANISMS BETWEEN WEIGHT LOSS-SENSITIVE AND -RESISTANT BLOOD PRESSURE REDUCTION IN OBESE SUBJECTS. HYPERTENS RES. 2001;24:371–376.
- 50. HARTE AL, MCTERNAN PG, MCTERNAN CL, CROCKER J, STARCYNSKI J, BARNETT AH, MATYKA K, KUMAR S. INSULIN INCREASES ANGIOTENSINOGEN EXPRESSION IN HUMAN ABDOMINAL SUBCUTANEOUS ADIPOCYTES. DIABETES OBES METAB. 2003;5:462–467.
- 51. ENGELI S, SCHLING P, GORZELNIAK K, BOSCHMANN M, JANKE J, AILHAUD G, TEBOUL M, MASSIERA F, SHARMA AM. THE ADIPOSE-TISSUE RENIN-ANGIOTENSIN- ALDOSTERONE SYSTEM: ROLE IN THE METABOLIC SYNDROME? INT J BIOCHEM CELL BIOL. 2003;35:807–825.
- 52. ANDRONICO G, COTTONE S, MANGANO MT, FERRARO-MORTELLARO R, BAIARDI G, GRASSI N, FERRARA L, MULE G, CERASOLA G. INSULIN, RENIN-ALDOSTERONE SYSTEM AND BLOOD PRESSURE IN OBESE PEOPLE. INT J OBES RELAT METAB DISORD. 2001;25:239 –242.
- 53. GOODFRIEND TL, CALHOUN DA. RESISTANT HYPERTENSION, OBESITY, SLEEP APNEA, AND ALDOSTERONE: THEORY AND THERAPY. HYPERTENSION. 2004;43: 518–524.134.
- 54. GOODFRIEND TL, BALL DL, EGAN BM, CAMPBELL WB, NITHIPATIKOM K. EPOXY-KETO DERIVATIVE OF LINOLEIC ACID STIMULATES ALDOSTERONE SECRETION.HYPERTENSION. 2004;43:358 –363.
- 55. REISIN E, FROHLICH ED, MESSERLI FH, DRESLINSKI GR, DUNN FG, JONES MM, BATSON HM JR. CARDIOVASCULAR CHANGES AFTER WEIGHT REDUCTION IN OBESITY HYPERTENSION. ANN INTERN MED. 1983;98:315–319.
- 56. TUCK ML, SOWERS J, DORNFELD L, KLEDZIK G, MAXWELL M. THE EFFECT OF WEIGHT REDUCTION ON BLOOD PRESSURE, PLASMA RENIN ACTIVITY, AND PLASMA ALDOSTERONE LEVELS IN OBESE PATIENTS. N ENGL J MED. 1981;304:930 –933.
- 57. SLEEP-RELATED BREATHING DISORDERS IN ADULTS: RECOMMENDATIONS FOR SYNDROME DEFINITION AND MEASUREMENT TECHNIQUES IN CLINICAL RESEARCH: THE REPORT OF AN AMERICAN ACADEMY OF SLEEP MEDICINE TASK FORCE.SLEEP. 1999;22:667–689.

- 58. POIRIER P, GILES TD, BRAY GA, HONG Y, STERN JS, PI-SUNYER FX, ECKEL RH; AMERICAN HEART ASSOCIATION; OBESITY COMMITTEE OF THE COUNCIL ON NUTRITION, PHYSICAL ACTIVITY, AND METABOLISM. OBESITY AND CARDIOVASCULAR DISEASE: PATHOPHYSIOLOGY, EVALUATION, AND EFFECT OF WEIGHT LOSS: AN UPDATE OF THE 1997 AMERICAN HEART ASSOCIATION SCIENTIFIC STATEMENT ON OBESITY AND HEART DISEASE FROM THE OBESITY COMMITTEE OF THE COUNCIL ON NUTRITION, PHYSICAL ACTIVITY, AND METABOLISM. CIRCULATION. 2006;113: 898–918.
- 59. KASPER EK, HRUBAN RH, BAUGHMAN KL. CARDIOMYOPATHY OF OBESITY: A CLINICOPATHOLOGIC EVALUATION OF 43 OBESE PATIENTS WITH HEART FAILURE. AM J CARDIOL. 1992;70:921–924.
- 60. ALPERT MA, FRALEY MA, BIRCHEM JA, SENKOTTAIYAN N. MANAGEMENT OF OBESITY CARDIOMYOPATHY. EXPERT REV CARDIOVASC THER. 2005;3:225–230.
- MESSERLI FH. CARDIOPATHY OF OBESITY: A NOT-SO-VICTORIAN DISEASE. N ENGL J MED. 1986;314:378 –380.
- 62. KU CS, LIN SL, WANG DJ, CHANG SK, LEE WJ. LEFT VENTRICULAR FILLING IN YOUNG NORMOTENSIVE OBESE ADULTS. AM J CARDIOL. 1994;73:613–615.
- 63. ASHRAFIAN H, LE ROUX CW, DARZI A, ATHANASIOU T. EFFECTS OF BARIATRIC SURGERY ON CARDIOVASCULAR FUNCTION. CIRCULATION. 2008;118:2091–2102
- 64. SACKS HS, FAIN JN. HUMAN EPICARDIAL ADIPOSE TISSUE: A REVIEW. AM HEART J. 2007;153:907–917.
- 65. IACOBELLIS G, CORRADI D, SHARMA AM. EPICARDIAL ADIPOSE TISSUE: ANATOMIC, BIOMOLECULAR AND CLINICAL RELATIONSHIPS WITH THE HEART. NATCLIN PRACT CARDIOVASC MED. 2005;2:536 –543.
- 66. IACOBELLIS G, BARBARO G. THE DOUBLE ROLE OF EPICARDIAL ADIPOSE TISSUE AS PRO- AND ANTI-INFLAMMATORY ORGAN. HORM METAB RES. 2008;40:442–445.
- 67. VELA D, BUJA LM, MADJID M, BURKE A, NAGHAVI M, WILLERSON JT, CASSCELLS SW, LITOVSKY S. THE ROLE OF PERIADVENTITIAL FAT IN ATHEROSCLEROSIS. ARCH PATHOL LAB MED. 2007;131:481–487.
- 68. BAKER AR, SILVA NF, QUINN DW, HARTE AL, PAGANO D, BONSER RS, KUMAR S, MCTERNAN PG. HUMAN EPICARDIAL ADIPOSE TISSUE

- EXPRESSES A PATHOGENIC PROFILE OF ADIPOCYTOKINES IN PATIENTS WITH CARDIOVASCULAR DISEASE. CARDIOVASC DIABETOL. 2006: 5:1.
- 69. MACMAHON SW, WILCKEN DE, MACDONALD GJ. THE EFFECT OF WEIGHT REDUCTION ON LEFT VENTRICULAR MASS: A RANDOMIZED CONTROLLED TRIAL IN YOUNG, OVERWEIGHT HYPERTENSIVE PATIENTS. N ENGL J MED. 1986;314: 334–339.
- 70. ALPERT MA, LAMBERT CR, TERRY BE, COHEN MV, MULEKAR M, MASSEY CV, HASHIMI MW, PANAYIOTOU H, MUKERJI V. EFFECT OF WEIGHT LOSS ON LEFT VENTRICULAR DIASTOLIC FILLING IN MORBID OBESITY. AM J CARDIOL. 1995; 76:1198 –1201.
- 71. ALPERT MA, ET AL.. FACTORS INFLUENCING LEFT VENTRICULAR SYSTOLIC FUNCTION IN NONHYPERTENSIVE MORBIDLY OBESE PATIENTS, AND EFFECT OF WEIGHT LOSS INDUCED BY GASTROPLASTY. AM J CARDIOL. 1993;71:733–737.
- 72. MCCLOSKEY CA, RAMANI GV, MATHIER MA, SCHAUER PR, EID GM, MATTAR SG, COURCOULAS AP, RAMANATHAN R. BARIATRIC SURGERY IMPROVES CARDIAC FUNCTION IN MORBIDLY OBESE PATIENTS WITH SEVERE CARDIOMYOPATHY. SURG OBES RELAT DIS. 2007;3:503–507.
- 73. RISTOW B, RABKIN J, HAEUSSLEIN E. IMPROVEMENT IN DILATED CARDIOMYOPATHY AFTER BARIATRIC SURGERY. J CARD FAIL. 2008;14:198